CLINICAL TRIAL: NCT05223504
Title: WARD-Home - Continuous Monitoring of Vital Parameters for Early Detection of Complications in Patients Discharged After Acute Medical Hospitalization
Brief Title: WARD-Home - Continuous Monitoring of Vital Parameters After Discharge
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Technical University of Denmark (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Vibeke Eriksen, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: WARD-Home feasibility
Record Dates: First submitted 2022-01-20; First posted 2022-02-04 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Vital Sign; Clinical Deterioration
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed patients: Adult patients (≥18 years) admitted with an acute medical disease and who are scheduled for discharge to their own homes within five days from inclusion.
  Interventions: Device: Continuously monitoring

INTERVENTIONS:
Device: Continuously monitoring — Included patients are monitored with WARD equipment during the last part of hospitalization and the first days after discharge. Monitoring will last for a maximum of eight days.

SUMMARY:
The current pilot study aims to investigate the feasibility of wireless, continuous monitoring of patients in the days around discharge after an acute medical hospitalization, as well as occurrence of deviating vital signs in this patient group.

DETAILED DESCRIPTION:
The healthcare system is challenged by an aging patient population with chronic diseases, and acute admissions must be housed in hospitals with fewer beds and less staff resources. This increases the need for earlier discharge and for treatment shifted to the patients' own home. Furthermore, the transition from the hospital to the home setting is one of potential hazard, due to the lack of observation and intervention possibilities.

This pilot study aims to investigate the feasibility of wireless, continuous monitoring of patients in the days around discharge after an acute medical hospitalization, as well as occurrence of deviating vital signs i in the patients' own homes during the first days after discharge.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years) Admitted with an acute medical disease and scheduled for discharge to their own homes within five days from inclusion.

Exclusion Criteria:

* Allergy to plaster, plastic, or silicone.
* A pacemaker or Implantable Cardioverter Defibrillator (ICD) device.
* If the patient was deemed not able to open the front door when visited by the investigator.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with an acute medical disease at Bispebjerg Hospital and scheduled for discharge to their own homes within five days from inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Duration of data collection from the Lifetouch patch | Up to 8 days of monitoring

SECONDARY OUTCOMES:
Duration of complete peripheral saturation data | Up to 8 days of monitoring
Duration of complete blood pressure data | Up to 8 days of monitoring
Cummulated duration of desaturation | Up to 8 days of monitoring
  Peripheral saturation below 88% and 85%
Number of events with SpO2 < 88% in at least 10 consecutive minutes | Up to 8 days of monitoring
Number of events with SpO2 < 85% in at least 5 consecutive minutes | Up to 8 days of monitoring
Number of deviating vital parameters in accordance to defined microevents | Up to 8 days of monitoring

OTHER OUTCOMES:
Re-admission and cause of re-admission within 30-days | 30-days follow up

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke R Eriksen, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Bispebjerg and Frederiksberg hospital, København NV, Region H, Denmark

IPD SHARING:
Plan to Share IPD: No